CLINICAL TRIAL: NCT06844968
Title: Multi-Faced Optimization of Sports Training Focused on Training Status Energy and Muscle Adaptation to Effort
Brief Title: The Effect of a 2000-m Ergometer Test on Training Status Indicators and the Muscle Adaptation in Rowers
Acronym: ETTETTSIAMAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Rowers 2024; RPW/8857/2024 (Other: Ministry of Sport and Tourism)
Record Dates: First submitted 2025-01-09; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Exhaustion - Physiological
Keywords: rowers; EPO; VEGF; hypoxanthine; glycogen; athletes
MeSH Terms: interventions — Physical Exertion

STUDY DESIGN:
Intervention Model Description: A group of rowers subjected to an efford on a rowing ergometer. The examined rowers group will be subjected to an effort on a rowing ergometer, consisting of covering a designated distance in the shortest possible time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical effort (Other): The effort on the rowing ergometer, based on swimming a specified distance in the shortest possible time.
  Interventions: Other: Physical effort

INTERVENTIONS:
Other: Physical effort — The examined rowers will be subjected to an effort on a rowing ergometer, consisting of covering a designated distance in the shortest possible time.
  Other Names: Rowing ergometer test

SUMMARY:
Intense physical exercise can lead to micro-damage to tissues and activation of inflammatory processes, the body's natural response to exercise-related metabolic stress. Monitoring inflammation and fatigue will enable the observation of athletes in terms of post-exercise regeneration and muscle adaptation to physical effort. The obtained results will allow for estimating the level of fatigue, minimizing the risk of injury, and will show the rate of post-exercise regeneration or its absence.

DETAILED DESCRIPTION:
The study will involve 40 members of the Polish Youth Rowing Team, both sexes, aged 19-23. The study will be held on three dates related to the specifics of the athletes' training cycle, i.e. in the preparatory period (March), the competition period (June), and the detraining period (November). The participants will perform an intensive exercise test on a rowing ergometer (manufacturer: Concept II, USA), covering a distance of 2,000 meters in the shortest possible time. The study will involve 40 members of the Polish Youth Rowing Team, both sexes, aged 19-23. Each time, before starting the exercise test, a non-invasive anthropometric analysis will be performed using the TANITA MC-780MA body composition analyzer (tanita Japan), to determine the body composition: percentage of body fat, body fat mass, lean tissue mass, muscle mass, body water and body mass index (BMI). On the three indicated dates, before and after the stress test, capillary blood (ear lobe) from the cubital vein will be collected from the participants. Using immunoenzymatic ELISA tests, the following will be determined: EPO (erythropoietin), VEGF (vascular endothelial growth factor), CRP (C-reactive protein), glycogen, hypoxanthine (Hx). Glucose level will be determined using an Accu-Chek Active glucometer (Roche, Germany).

ELIGIBILITY:
Inclusion Criteria:

* members of the Polish Youth Rowing Team - competitors officially called up to the Polish national rowing team,
* no musculoskeletal injuries that would prevent them from performing the exercise test,
* written consent of the competitor to participate in the study.

Exclusion Criteria:

* anti-inflammatory drugs, other supplements in the last 3 months before starting the study,
* failure to complete the test,
* current injury, post-traumatic condition, illness,
* lack of informed consent of the athlete.

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
EPO (erythropoietin) level | Immediately before the ergometer test, immediately after and 3 hours after the test
  Immunoenzymatic assay method using a diagnostic ELISA Kit
VEGF (vascular endothelial growth factor) level | Immediately before the ergometer test, immediately after and 3 hours after the test
  Immunoenzymatic assay method using a diagnostic ELISA Kit
Hypoxanthine (Hx) level | Immediately before the ergometer test, immediately after and 3 hours after the test
  Immunoenzymatic assay method using a diagnostic ELISA Kit
Glycogen level | Immediately before the ergometer test, immediately after and 3 hours after the test
  Immunoenzymatic assay method using a diagnostic ELISA Kit
Glucose level | Immediately before the ergometer test, immediately after and 3 hours after the test
  Using an Accu-Chek Active glucometer (Roche, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kasperska, PhD, Principal Investigator — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;
Locations (1):
- Poznań University of Physical Education, Faculty of Physical Culture in Gorzów Wielkopolski, Gorzów Wielkopolski, Polska, Poland

IPD SHARING:
Plan to Share IPD: No